CLINICAL TRIAL: NCT01589809
Title: Pharmacodynamic Studies of a Histone Deacetylase Inhibitor in Friedreich's Ataxia
Brief Title: Effect of Nicotinamide in Friedreich's Ataxia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR01849
Record Dates: First submitted 2012-02-20; First posted 2012-05-02 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-01

CONDITIONS: Neurodegenerative Disorders
Keywords: Congenital, familial and genetic disorders; Nervous System Diseases
MeSH Terms: conditions — Neurodegenerative Diseases; Genetic Diseases, Inborn; Nervous System Diseases | interventions — Niacinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nicotinamide (Experimental): Comparison is made within-subjects to different doses and no treatment
  Interventions: Drug: nicotinamide

INTERVENTIONS:
Drug: nicotinamide — dose-escalation, 2-8 grams, oral
  Other Names: Vitamin B3

SUMMARY:
The purpose of the interventional study is to determine whether Nicotinamide is effective at upregulating the Frataxin (FXN) gene in patients with Friedreich's ataxia (FRDA) where this gene is abnormally 'switched off'.

The purpose of the non-interventional study is to investigate the use of novel, highly-sensitive technology to capture clinical deficit and measure subtle changes in the activities of daily living and to correlate functional changes to levels of expression of Frataxin protein and the epigenetic structure of the Frataxin gene over a 9-12 month period without nicotinamide. Healthy volunteers will be included as comparators in this part of the study.

DETAILED DESCRIPTION:
Friedreich's ataxia (FRDA) is caused by a GAA repeat expansion in the Frataxin gene causing its repression which resembles the archetypal epigenetic phenomenon of Position Effect Variegation and hence can be modulated by chromatin modifiers The investigators have now confirmed that a similar form of silencing occurs in cells from FRDA patients. Based on these findings histone deacetylase (HDAC) inhibitors which can overcome such silencing have been identified. The investigators have extended this result by showing that the classical Class III HDAC inhibitor, nicotinamide, can relieve silencing in cells from patients. Nicotinamide is a vitamin and a registered drug and has been previously administered to humans with no significant ill effects.

In the interventional study, the investigators will perform pharmacodynamic studies on nicotinamide in humans with FRDA to investigate whether the investigators can upregulate Frataxin and if so, to determine an optimum dosing regimen. Nicotinamide will be administered orally following a standard drug escalation regimen and blood samples taken to measure Frataxin level and chromatin structure of the Frataxin gene. The end-point of the study is to achieve significant upregulation of Frataxin in patients providing a potential therapy for this currently untreatable condition.

In the non-interventional study, we will investigate the use of novel, highly-sensitive technology to capture clinical deficit and measure subtle changes in the activities of daily living and correlate functional changes to levels of expression of Frataxin protein and the epigenetic structure of the Frataxin gene over a 9-12 month period without nicotinamide. Healthy volunteers as comparators will be included in this part of the study. HVs will undergo the same assessments as participants with Friedreich ataxia once.

ELIGIBILITY:
Inclusion Criteria for the interventional study

1. Participants must have a molecular genetic diagnosis of FRDA, consisting of a GAA-repeat expansion on both alleles of the FXN gene.
2. Participants must be over the age of 18 years living in the UK and registered with a GP.
3. Participants must provide informed consent. If written consent is not possible due to physical incapacity, written consent on behalf of the participant will be sought from the participant's relatives or carer.
4. A female participant is eligible to participate if she is of:

Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol <40 pg/ml (<140 pmol/L) is confirmatory].

Child-bearing potential and agrees to use one of the following contraception methods:

True abstinence: When this is in line with the preferred and usual lifestyle of the participant. [Periodic abstinence (e.g.,calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception].

Contraceptive Methods with a Failure Rate of < 1%:

* Oral contraceptive, either combined or progestogen alone;
* Injectable progestogen;
* Implants of levonorgestrel;
* Estrogenic vaginal ring;
* Percutaneous contraceptive patches; -
* Intrauterine device (IUD) or intrauterine system (IUS) that meets the <1% failure rate as stated in the product label;
* Male partner(s) sterilisation (vasectomy with documentation of azoospermia) prior to the female participants entry into the study;
* Double barrier method: condom and occlusive cap (diaphragm or cervical/vault caps) plus vaginal spermicidal agent (foam/gel/film/cream/suppository).

Exclusion Criteria for the interventional study

1. Participants with significant clinical dysphagia.
2. Participants taking Sodium Valproate or any other known histone deacetylase inhibitor.
3. Participants taking part in another interventional clinical trial or who have done so within 30 days before screening.
4. Participants known to be positive for human immunodeficiency virus (HIV).
5. Participants with any additional medical condition or illness that, in the opinion of the CI would interfere with study compliance and/or impair the participants ability to participate or complete the study. Concurrent diseases or conditions that may interfere with study participation or safety include liver disease, bleeding disorders, arrhythmias, organ transplant, organ failure, current neoplasm, poorly controlled diabetes mellitus, poorly controlled hypertension, clinically significant haematological or biochemical abnormality.
6. Patients with a history of substance abuse (e.g. alcohol or drug abuse) within the previous 6 months before enrolment.
7. Participants with a history of severe allergies.
8. Female participants who are lactating or pregnant (positive pre-randomisation serum pregnancy test) or plan to become pregnant during the study.
9. Hypersensitivity to Nicobion (nicotinamide) or any of the excipients in this preparation
10. Liver function tests outside the normal range: aspartate aminotransferase (AST), alanine aminotransferase (ALT), bilirubin which in the opinion of the CI would put the participants safety at risk.

Inclusion Criteria for the non-interventional study

1. Up to 20 participants must have a molecular genetic diagnosis of FRDA, consisting of a GAA-repeat expansion on both alleles of the FXN gene.

   Up to 20 participants must be HV.
2. Participants are over the age of 18 years, living in the UK and registered with a GP.
3. Participants must provide informed consent. If written consent is not possible due to physical incapacity, written consent on behalf of the participant will be sought from the participant's relatives or carer.
4. Women of child-bearing potential must have a negative urine pregnancy test.

Exclusion Criteria for the non-interventional study

1. Contraindications to MRI including, but not limited to: intracranial aneurism clips (except Sugita), history of metal lathe work or possibility of intra-orbital metal fragments, pacemakers and non-MR compatible heart valves or other non-MR compatible implants, history of claustrophobia or participant feels unable to lie still on their back for a period of 60-90mins in the fMRI scanner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-06; Primary Completion 2015-06 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Significant upregulation of Frataxin (FXN) in patients with Friedrich ataxia using an antibody dipstick assay (interventional part) | Daily administration up to 9 weeks
  Low levels of Frataxin (FXN) (<30% of normal) cause Friedrich ataxia. The trial will determine the effect of oral nicotinamide in upregulating FXN. Therefore the primary outcome is upregulation of Frataxin levels above baseline. This will be measured using an antibody dipstick assay (Mitosciences) and chromatin immunoprecipitation studies.

SECONDARY OUTCOMES:
Assessment of impact on clinical phenotype using the SARA scale to measure degree of ataxia (interventional part of the study) | Daily administration up to 9 weeks
  Assessment of impact on clinical phenotype using the SARA scale to measure degree of ataxia
Use of novel highly-sensitive technology to capture clinical deficit (non-interventional part) | 6-9 months
  Investigate the use of novel, highly-sensitive technology to capture clinical deficit and measure subtle changes in the activities of daily living over a 6-9 month period without nicotinamide.
Correlate functional changes to levels of expression of Frataxin protein and the epigenetic structure of the Frataxin gene over a 6-9 month period without nicotinamide (non-interventional part). | 6-9 months
  Correlate functional changes to levels of expression of Frataxin protein and the epigenetic structure of the Frataxin gene over a 6-9 month period without nicotinamide (non-interventional part).
Assessment of additional FRDA biomarkers using gene expression profiling (interventional study). | Daily administration up to 9 weeks
  Assessment of additional FRDA biomarkers using gene expression profiling (interventional study).
Chromatin immunoprecipitation (interventional study) | Daily administration up to 9 weeks
  Further assessment of efficacy by means of chromatin immunoprecipitation to look for epigenetic changes at the Frataxin locus compatible with transcriptional upregulation. Such information might also be useful in identifying patients more likely to respond to this therapy by upregulating FXN (interventional study).
Determine the safety and tolerability of nicotinamide in FRDA patients (interventional study). | Daily administration up to 9 weeks.
  Determine the safety and tolerability of nicotinamide in FRDA patients (interventional study).

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Libri, Dr, Principal Investigator — Imperial College London; Paola Giunti, Dr, Principal Investigator — NHNN, 02034483153
Locations (2):
- United Kingdom (2):
  - NIHR/Wellcome Trust Imperial CRF, London, Hammersmith
  - National Hospital for Neurology and Neurosurgery, London

REFERENCES:
- [Derived] Libri V, Yandim C, Athanasopoulos S, Loyse N, Natisvili T, Law PP, Chan PK, Mohammad T, Mauri M, Tam KT, Leiper J, Piper S, Ramesh A, Parkinson MH, Huson L, Giunti P, Festenstein R. Epigenetic and neurological effects and safety of high-dose nicotinamide in patients with Friedreich's ataxia: an exploratory, open-label, dose-escalation study. Lancet. 2014 Aug 9;384(9942):504-13. doi: 10.1016/S0140-6736(14)60382-2. Epub 2014 Apr 30. PMID 24794816